CLINICAL TRIAL: NCT06768242
Title: Inter- and Intra-fraction Fiducial Position Reproducibility in End-exhalation Breath Hold for Ethos Liver Radiotherapy - Part of the Modern Art Study
Brief Title: Part of the Modern Art Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Alejandra Mendez Romero, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL86070.078.24
Record Dates: First submitted 2024-12-24; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: HCC - Hepatocellular Carcinoma; Liver Metastases
Keywords: HCC - Hepatocellular Carcinoma; Stereotactic body radiation therapy; Breath hold; Liver metastases
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cone beam CT (Experimental): Single-arm study
  Interventions: Radiation: Cone beam CT

INTERVENTIONS:
Radiation: Cone beam CT — Each patient will undergo three cone beam CTs per session, and a total of three sessions.

SUMMARY:
One of the possible treatments for patients with liver tumours (hepatocellular carcinoma (HCC) or liver metastases) at the Erasmus MC is stereotactic body radiation therapy (SBRT) on the Cyberknife. To spare the organs at risk, suboptimal coverage of the planning target volume is sometimes accepted. The Ethos treatment system is equipped with a novel cone-beam CT (CBCT), which provides higher quality images. This makes it possible to consider online adaptive radiotherapy with daily plan adaptation, potentially leading to a higher dose on the tumour whilst sparing the surrounding healthy tissue more.

Liver tumours move with the breathing motion. On the CyberKnife, a tracking technology is used to keep track of the tumour, but this is not available on the Ethos. Because of this, breath holds will be used for breathing management, but appropriate safety margins need to be established under the new treatment conditions. The aim of this study is to determine the reproducibility of the tumour position for each breath hold within a treatment fraction, and also between treatment fractions, which is a crucial component in the establishment of appropriate safety margins.

DETAILED DESCRIPTION:
Rationale:

One of the possible treatments for patients with liver tumours (hepatocellular carcinoma (HCC) or liver metastases) at the Erasmus MC is stereotactic body radiation therapy (SBRT) on the Cyberknife. To spare the organs at risk, suboptimal coverage of the planning target volume is sometimes accepted on the Cyberknife. The Ethos therapy linear accelerator is equipped with a novel cone-beam CT (CBCT), which provides higher quality images. This makes it possible to consider online adaptive radiotherapy with daily plan adaptation, potentially leading to a higher dose on the tumour whilst sparing the surrounding healthy tissue more.

Objectives:

To determine inter- and intra-fraction fiducial and patient position reproducibility in order to determine appropriate safety margins for liver SBRT treatment on Ethos.

Study design:

A prospective, single arm cohort study.

Study population:

Ten patients, either with liver metastases (all ages), or age ≥ 65 years with HCC, who are referred to the department of Radiotherapy for SBRT, able to comply with breath-hold requirements and not eligible for liver transplantation or curative surgery.

Intervention:

Nine CBCTs for each patient in end-exhalation breath hold on t Main study parameters/endpoints: The primary parameters are inter- and intra-fraction fiducial position reproducibility on the Ethos.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Patient discussed in multidisciplinary tumor board;
* Patient diagnosed with liver metastases and referred to the dept. of Radiotherapy for SBRT OR patient ≥65 years, diagnosed with HCC and referred to the dept. of Radiotherapy for SBRT;
* Able to comply with breath-hold requirements.

Exclusion Criteria:

* Eligibility for surgery, ablation or liver transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Intrafraction fiducial position reproducibility | Before or after three radiotherapy sessions over the course of treatment.
  The translation in mm in three directions (craniocaudal, left-right and anterior-posterior) of each of the fiducials in the second and third cone beam CT, compared to the first cone beam CT of each session.
Interfraction fiducial position reproducibility | Before or after three radiotherapy sessions over the course of treatment.
  The translation in mm in three directions (craniocaudal, left-right and anterior-posterior) of each of the fiducials in each of the imaging sessions, compared to the planning CT that was made before the start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Méndez Romero, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No